CLINICAL TRIAL: NCT01085903
Title: Identifying and Treating Arousal Related Deficits in Neglect and Dysphagia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 110644; R21HD055677 (NIH)
Record Dates: First submitted 2010-03-09; First posted 2010-03-12 (Estimated); Results first posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Spatial Neglect; Dysphagia
Keywords: Spatial Neglect; Dysphagia; Arousal; Modafinil; Stroke
MeSH Terms: conditions — Deglutition Disorders; Stroke | interventions — Modafinil; Noble Gases; BaseLine dental cement

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- normal subjects (Active Comparator): Normal subjects are persons without stroke who receive baseline, CPS, Post CPS and Follow up interventions.
  Interventions: Behavioral: Baseline; Behavioral: CPS; Behavioral: Post CPS; Behavioral: Follow up
- stroke subjects (Active Comparator): Stroke subjects are persons who have had a stroke affecting the right hemisphere and are subject to neglect or dysphagia who receive modafinil, placebo, baseline, CPS, Post CPS and Follow up interventions.
  Interventions: Drug: Modafinil; Drug: Placebo; Behavioral: Baseline; Behavioral: CPS; Behavioral: Post CPS; Behavioral: Follow up

INTERVENTIONS:
Drug: Modafinil — 200 mg once daily with morning meal for three days administered only to stroke patients
  Other Names: Provigil
  Arms: stroke subjects
Drug: Placebo — Subjects will receive a placebo designed to look like 200 mg dose of modafinil. The dose will be taken once daily with the morning meal for three days and will only be administered to stroke patients
  Other Names: inert
  Arms: stroke subjects
Behavioral: Baseline — Observations made at baseline before any intervention
  Other Names: baseline observation
Behavioral: CPS — Submerging each participant's foot into ice water (36-44 F) for 50 seconds.
  Other Names: cold pressor stimulation
Behavioral: Post CPS — 20 minutes following the CPS condition.
  Other Names: post cold pressor stimulation
Behavioral: Follow up — Follow up testing occurred at 3 months
  Other Names: three month follow up

SUMMARY:
The purpose of this study is to examine how stroke can alter arousal, alertness, neglect and dysphagia, and whether a medication, modafinil, can improve arousal.

DETAILED DESCRIPTION:
Neglect and dysphagia are two of the most problematic behavioral disorders encountered in stroke rehabilitation with 300,000 patients affected annually in the US. Both disorders impede progress in therapy and both lead to costly medical complications, like falls which are associated with neglect and aspiration pneumonia and malnutrition which are associated with dysphagia. No widely accepted pharmacological treatment exists for either disorder.

A new direction of this application is to view neglect and dysphagia as different disorders that share a common deficit in magnitude estimation (ME). ME refers to one's ability to perceive the intensity of sensory stimulation. Deficits in ME explain how much of a stimulus is neglected by stroke patients. Sensory deficits are also known to produce dysphagia. Perceptual deficits influence how patients response to stimuli like failing to act on all stimuli present (neglect) and failing to generate swallowing reflexes sufficient for normal bolus flow (dysphagia).

We know from previous work that ME is altered by change in cortical arousal following stroke (decreased or hypoarousal). Hypoarousal is evidenced by objective and subjective post-stroke fatigue and daytime sleepiness which occurs in 50% of stroke patients and can persist chronically. Increasing arousal could potentially reverse the perceptual deficits associated with hypoarousal and improve neglect and dysphagia. This proposal manipulates arousal in two ways. Cold pressor stimulation (CPS), immersing the foot in cold water for 50 seconds, is used to increase arousal and reverse neglect and dysphagia temporarily. A brief, 3-day trial of modafinil (Provigil) versus placebo is then used in stroke patients to learn if a positive response to cold-pressor stimulation can predicts patients who respond positively to modafinil.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Willingness to complete study procedures
* Ability to comprehend and sign informed consent
* Evidence of unilateral, ischemic stroke based on:

  * Neuroimaging (clinically obtained imaging studies showing evidence of stroke)

    * Acceptable categories of stroke include:
    * Unilateral ischemic stroke
    * Atherothrombotic stroke
    * Cardioembolic stroke
    * Lacunar stroke >1.5 cm
    * Chronic stable, unilateral hemorrhagic stroke
* Or Behavioral evidence of stroke including:

  * Hemiplegia
  * Unilateral sensory impairment
  * Localized higher cortical dysfunction (e.g. neglect,dysphagia, apraxia)

Exclusion Criteria:

* Cardiac valvular disease
* Left heart hypertrophy
* Poorly controlled hypertension
* Active variant angina
* Pre-menopausal women capable of having children, including those using active contraception (precaution for study medication and not applicable to normal subjects)
* Severe renal or hepatic disease
* History of psychosis or substance abuse
* Patients on other Central Nervous System (CNS) stimulants, dopamine agonists or antagonists (antipsychotics)
* Severe speech comprehension deficit and/or inability to communicate responses
* Allergies that could put the research subject at risk during the course of the study
* Cannot speak English
* Active cerebral neurologic disease other than stroke such as multiple sclerosis or Alzheimer's Disease
* Active psychiatric illness except past history of treated depression or anxiety disorders
* For persons needing an MRI - standard MRI exclusion criteria (cardiac pacemaker or defibrillator, artificial heart valves, metallic aneurysm clips eye or ear implants, implanted insulin or infusion pumps, battery activated stimulators, and history of claustrophobia)
* Concomitant medications excluded: Based on recommendations of manufacturer, the following concomitant medications are excluded: Tricyclic antidepressants and Monoamine oxidase (MAO) inhibitors. Any other CNS stimulation producing medications. Antifungal agents Itraconazole or Ketoconazole as plasma concentrations of modafinil may be increased.
* Stroke patients will be excluded from the modafinil trial if they cannot swallow a capsule.
* Stroke patients are excluded if they are able to become pregnant
* Any other criteria that the PI or study physicians feel would put the volunteer's health at risk during the course of the study

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Mennemeier, PhD, Principal Investigator — University of Arkansas; Gary McCullough, PhD, Principal Investigator — University of Central Arkansas
Locations (2):
- United States (2):
  - Conway Regional Rehabilitation Hospital, Conway, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Subjects Baseline: Normal subjects are persons without stroke who receive baseline, Cold Pressor Stimulation (CPS), Post CPS and Follow up interventions.
  Baseline: Observations made at baseline before any intervention
  CPS: Submerging each participant's foot into ice water (36-44 F) for 50 seconds.
  Post CPS: 20 minutes following the CPS condition.
- Stroke Subjects: Placebo Then Modafinil; Stroke Subjects: Modafinil Then Placebo: Denotes sequence Modafinil: 200 mg once daily with morning meal for three days administered only to stroke patients
  Placebo: Subjects will receive a placebo designed to look like 200 mg dose of modafinil. The dose will be taken once daily with the morning meal for three days and will only be administered to stroke patients
  Baseline: Observations made at baseline before any intervention
  CPS: Submerging each participant's foot into ice water (36-44 F) for 50 seconds.
  Post CPS: 20 minutes following the CPS condition.
Period: Overall Study
Arm/Group | Normal Subjects Baseline | Stroke Subjects: Placebo Then Modafinil | Stroke Subjects: Modafinil Then Placebo
Started | 21 | 4 | 3
Completed | 21 | 4 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Stroke Subjects: Stroke subjects are persons who have had a stroke affecting the right hemisphere and are subject to neglect or dysphagia who receive baseline, CPS, and Post CPS and then are randomized to modafinil or placebo.
  Baseline: Observations made at baseline before any intervention
  CPS: Submerging each participant's foot into ice water (36-44 F) for 50 seconds.
  Post CPS: 20 minutes following the CPS condition. Modafinil: 200 mg once daily with morning meal for three days administered only to stroke patients
  Placebo: Subjects will receive a placebo designed to look like 200 mg dose of modafinil. The dose will be taken once daily with the morning meal for three days and will only be administered to stroke patients
- Total: Total of all reporting groups
Arm/Group | Normal Subjects | Stroke Subjects | Total
Number analyzed (Participants) | 21 | 7 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.286 (21.462) | 71.429 (9.914) | 58.2 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 13 | 4 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 18 | 6 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: P50 Percent Habituation Score
Description: This is an electrophysiological measure of arousal - a percent change in the P50 evoked response potential amplitudes with a 250 ms inter stimulus interval. The difference score is calculated as CPS - baseline and as modafinil - placebo (stroke subjects only).
Time Frame: baseline and after three days of intervention
Measure: Mean (Standard Deviation); unit: percentage of change in amplitude
Groups:
- Normal Subjects: Baseline vs CPS: Normal subjects are persons without stroke who receive baseline, CPS, Post CPS and Follow up interventions.
  Baseline: Observations made at baseline before any intervention
  CPS: Submerging each participant's foot into ice water (36-44 F) for 50 seconds.
- Stroke Subjects: Baseline vs CPS: Stroke subjects are persons who have had a stroke affecting the right hemisphere and are subject to neglect or dysphagia who receive modafinil, placebo, baseline, CPS, Post CPS and Follow up interventions.
  Baseline: Observations made at baseline before any intervention
  CPS: Submerging each participant's foot into ice water (36-44 F) for 50 seconds.
- Stroke Subjects: Modafinil: Modafinil: 200 mg once daily with morning meal for three days administered only to stroke patients
- Stroke Subjects: Placebo: Placebo: Subjects will receive a placebo designed to look like 200 mg dose of modafinil. The dose will be taken once daily with the morning meal for three days and will only be administered to stroke patients
- Stroke Subjects Placebo vs Modafinil: Placebo: Subjects will receive a placebo designed to look like 200 mg dose of modafinil. The dose will be taken once daily with the morning meal for three days and will only be administered to stroke patients
  Modafinil: 200 mg once daily with morning meal for three days administered only to stroke patients
Arm/Group | Normal Subjects: Baseline vs CPS | Stroke Subjects: Baseline vs CPS | Stroke Subjects: Modafinil | Stroke Subjects: Placebo | Stroke Subjects Placebo vs Modafinil
Number analyzed (Participants) | 21 | 7 | 7 | 7 | 7
percentage of change in amplitude | -44.12 (59.29) | -45.84 (228.09) | 113.63 (154.5) | 61.41 (102.5) | 52.223 (222.94)

2. Secondary Outcome: PVT Fastest 10 Percent of Reaction Times
Description: This is a behavioral measure of arousal - the fastest 10 percent of all cued reaction time trials. The difference score is calculated as CPS - baseline and as modafinil - placebo (stroke subjects only).
Time Frame: baseline and after three days of intervention
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Stroke Subjects: Baseline vs CPS: Stroke subjects are persons who have had a stroke affecting the right hemisphere and are subject to neglect or dysphagia who receive the baseline and CPS conditions and then are randomized to the placebo and modafinil interventions.
  Baseline: Observations made at baseline before any intervention
  CPS: Submerging each participant's foot into ice water (36-44 F) for 50 seconds.
- Stroke Subjects: Modafinil: Stroke subjects are persons who have had a stroke affecting the right hemisphere and are subject to neglect or dysphagia who receive the baseline and CPS conditions and then are randomized to the placebo and modafinil interventions.
  Modafinil: 200 mg once daily with morning meal for three days administered only to stroke patients
- Stroke Subjects: Placebo: Stroke subjects are persons who have had a stroke affecting the right hemisphere and are subject to neglect or dysphagia who receive the baseline and CPS conditions and then are randomized to the placebo and modafinil interventions.
  Placebo: Subjects will receive a placebo designed to look like 200 mg dose of modafinil. The dose will be taken once daily with the morning meal for three days and will only be administered to stroke patients
- Stroke Subjects Placebo vs Modafinil: Stroke subjects are persons who have had a stroke affecting the right hemisphere and are subject to neglect or dysphagia who receive the baseline and CPS conditions and then are randomized to the placebo and modafinil interventions.
  Modafinil: 200 mg once daily with morning meal for three days administered only to stroke patients
  Placebo: Subjects will receive a placebo designed to look like 200 mg dose of modafinil. The dose will be taken once daily with the morning meal for three days and will only be administered to stroke patients
Arm/Group | Normal Subjects: Baseline vs CPS | Stroke Subjects: Baseline vs CPS | Stroke Subjects: Modafinil | Stroke Subjects: Placebo | Stroke Subjects Placebo vs Modafinil
Number analyzed (Participants) | 21 | 7 | 7 | 7 | 7
milliseconds | -10.57 (21.66) | 20.57 (29.20) | 244.71 (186.62) | 235.64 (150.62) | 9.07 (38.73)

3. Secondary Outcome: Power Function Exponent for Oral Bolus Estimation
Description: This is a behavioral measure of sensation in the oral cavity. The power function exponent is equal to the slope of a regression equation relating bolus size to a person's estimate of that size. An exponent below one implies an underestimate of bolus size. The difference score is calculated as CPS - baseline and as modafinil - placebo (stroke subjects only).
Time Frame: baseline and after three days of intervention
Measure: Mean (Standard Deviation); unit: exponent
Groups:
- Stroke Subjects: Baseline vs CPS: Stroke subjects are persons who have had a stroke affecting the right hemisphere and are subject to neglect or dysphagia who receive baseline and CPS conditions before being randomized to placebo and modafinil.
  Baseline: Observations made at baseline before any intervention
  CPS: Submerging each participant's foot into ice water (36-44 F) for 50 seconds.
- Stroke Subjects: Modafinil: Stroke subjects are persons who have had a stroke affecting the right hemisphere and are subject to neglect or dysphagia who receive baseline and CPS conditions before being randomized to placebo and modafinil.
  Modafinil: 200 mg once daily with morning meal for three days administered only to stroke patients
- Stroke Subjects: Placebo: Stroke subjects are persons who have had a stroke affecting the right hemisphere and are subject to neglect or dysphagia who receive baseline and CPS conditions before being randomized to placebo and modafinil.
  Placebo: Subjects will receive a placebo designed to look like 200 mg dose of modafinil. The dose will be taken once daily with the morning meal for three days and will only be administered to stroke patients
- Stroke Subjects Placebo vs Modafinil: Stroke subjects are persons who have had a stroke affecting the right hemisphere and are subject to neglect or dysphagia who receive baseline and CPS conditions before being randomized to placebo and modafinil.
  Modafinil: 200 mg once daily with morning meal for three days administered only to stroke patients
  Placebo: Subjects will receive a placebo designed to look like 200 mg dose of modafinil. The dose will be taken once daily with the morning meal for three days and will only be administered to stroke patients
Arm/Group | Normal Subjects: Baseline vs CPS | Stroke Subjects: Baseline vs CPS | Stroke Subjects: Modafinil | Stroke Subjects: Placebo | Stroke Subjects Placebo vs Modafinil
Number analyzed (Participants) | 21 | 7 | 7 | 7 | 7
exponent | .014 (.113) | -.004 (.196) | .54 (.17) | .49 (.19) | .04 (.08)

4. Secondary Outcome: Time to Swallow Puree Food
Description: This is a behavioral measure of swallowing - the time it takes for pureed food to transition across a part of the throat. The difference score is calculated as CPS - placebo and as modafinil - placebo (for stroke subjects only).
Time Frame: baseline and after three days of intervention
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Normal Subjects: Baseline vs CPS: Normal subjects are persons without stroke who receive baseline and CPS conditions.
  Baseline: Observations made at baseline before any intervention
  CPS: Submerging each participant's foot into ice water (36-44 F) for 50 seconds.
- Stroke Subjects Placebo vs Modafinil: Stroke subjects are persons who have had a stroke affecting the right hemisphere and are subject to neglect or dysphagia who receive baseline and CPS conditions before being randomized to placebo and modafinil.
  Modafinil: 200 mg once daily with morning meal for three days administered only to stroke patients
  Placebo: Subjects will receive a placebo designed to look like 200 mg dose of modafinil. The dose will be taken once daily with the morning meal for three days and will only be administered to stroke patientseal for three days administered only to stroke patients
Arm/Group | Normal Subjects: Baseline vs CPS | Stroke Subjects: Baseline vs CPS | Stroke Subjects: Modafinil | Stroke Subjects: Placebo | Stroke Subjects Placebo vs Modafinil
Number analyzed (Participants) | 21 | 7 | 7 | 7 | 7
seconds | .029 (.121) | -.058 (.512) | .48 (1.05) | .12 (.11) | .36 (1.06)

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse Events were recorded in a cumulative fashion for stroke participants, and not according to the intervention received at the time of the event or according to the assigned intervention sequence.
Arm/Group | Normal Subjects | Stroke Subjects
Serious Adverse Events (participants affected / at risk) | 0/21 | 2/7
Other Adverse Events (participants affected / at risk) | 1/21 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Subjects (N=21) | Stroke Subjects (N=7)
stroke (Vascular disorders) | 0 | 1 — One participant had an additional stroke that was unrelated to the study
broken hip (Musculoskeletal and connective tissue disorders) | 0 | 1 — one participant broke a hip but this was not related to the study
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Subjects (N=21) | Stroke Subjects (N=7)
vasovagal response (Vascular disorders) | 1 (1) | 0 (0) — One normal subject had a vasovagal response during the swallowing evaluation
headache (Nervous system disorders) | 0 (0) | 2 (2) — headache with or without dizzyness
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) — rash with or without itchyness
difficulty sleeping (Nervous system disorders) | 0 (0) | 1 (1) — report of difficulty sleeping

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes